CLINICAL TRIAL: NCT03029845
Title: Propranolol for Treating Fibromyalgia Pain: Pilot Study
Brief Title: Propranolol for Treating Fibromyalgia Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The funding ended.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Akiko Okifuji, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00084875
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia Pain
MeSH Terms: interventions — propranolol mustard; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- propranolol 1 (Active Comparator): 20 mg propranolol twice a day
  Interventions: Drug: Propranolol 1
- propranolol 2 (Active Comparator): 10 mg propranolol twice a day
  Interventions: Drug: Propranolol 2
- Placebo (Placebo Comparator): Placebo twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol 1 — Participants will take 20 mg propranolol twice a day for 2 weeks
  Other Names: 20 mg propranolol
  Arms: propranolol 1
Drug: Propranolol 2 — Participants will take 10 mg propranolol twice a day for 2 weeks
  Other Names: 10 mg propranolol
  Arms: propranolol 2
Drug: Placebo — Participants will take placebo twice a day for 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study to evaluate the feasibility of using low dose propranolol for people with fibromyalgia.

DETAILED DESCRIPTION:
The main purpose of this study is to collect pilot feasibility study data for the use of low dose propranolol for helping treat fibromyalgia. The investigators plan to compare 20mg twice a day dosage of propranolol and 10mg twice a day dosage of propranolol to placebo. The design is a 3 arm, double blind randomized control trial. The investigators will also test ECG and respiratory assessment as a part of the safety screening and the feasible assessment of respiratory sinus arrhythmia.

Propranolol is not indicated to treat pain. However, the previous studies showed that low dose propranolol can re-regulate the adrenergic dysfunction and reduce pain in people with chronic musculoskeletal pain. However, the investigators are not aiming to develop a new indication of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Females with fibromyalgia (both meeting 1990 American College of Rheumatology (ACR) FMS criteria and 2010 ACR FMS criteria) age 18-65 with at least 1 year of symptoms and sedentary (exercising less than 120 min per week).

Exclusion Criteria:

* General Health Criteria:

  * Uncontrolled/unstable illnesses (physician diagnosed, self-report)
  * Pregnancy or planning to be pregnant in the next year
  * Having Asthma requiring medication treatment including inhaler
  * Type I diabetes or Type II diabetes requiring medical therapy that can lead to hypoglycemia
  * Having acute pain or neuropathic pain
  * Participation in exercise or psychological treatment studies in the past 2 years
  * Having known serious psychopathology: Psychosis, history of inpatient psychiatric admission in the past year, active suicidal intent, history of self-injurious behaviors in the past year, history of recreational IV drug use, substance abuse history in the past year)
* Cardiovascular Criteria:

  * Having known cardiovascular diseases (self-report, physician diagnosed)
  * Pacemaker
  * Bradycardia (resting heartrate of less than 55 bpm)
  * Resting diastolic BP < 55 mmHG or systolic BP<100 mmHG
  * ECG showing prolonged PR interval > .2 sec
  * ECG showing irregular PR interval
  * ECG showing incongruence between P wave and QRS
* Medication Criteria

  * Allergy or intolerance of beta blockers
  * Current use of the following drugs:

    * Antihypertensive drugs
    * Neuroleptics
    * Monoamine oxidase inhibitors
    * Tizanidine
    * Amphetamine-based medications
    * Bupropion
    * Mirtazapine
    * Tricyclics: daily dose greater than 75mg amitriptyline or equivalent
    * Benzodiazepine: daily dose greater than 5mg diazepam or equivalent
    * Asthmatic medicine, including inhaler
  * Participants may be included after minimum of 4 weeks of physician prescribed termination of these drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in self-reported measures of clinical pain using Fibromyalgia Impact Questionnaire - Revised (FIQ-R) | Pre (one week before start taking propranolol or placebo) and Post (immediately following the 14-day trial)
  Changes in clinical pain will be measured

SECONDARY OUTCOMES:
Change in self-reported measures of Fibromyalgia symptoms using Promis Fatigue | Pre (one week before start taking propranolol or placebo) and Post (immediately following the 14-day trial)
  Changes in fibromyalgia-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No